CLINICAL TRIAL: NCT06550219
Title: Evaluation of Nasal Non Invasive Ventilation Modalities in Management of Neonates With Respiratory Distress Using Lung Ultrasound
Brief Title: Evaluation of Nasal Non Invasive Ventilation in Management of Neonates With Respiratory Distress Using Lung Ultrasound
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Marwa Mohamed Farag, Assistant professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0108428
Record Dates: First submitted 2024-08-04; First posted 2024-08-12 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Preterm; Ventilator Lung; Newborn
Keywords: preterm infants; non-invasive ventilation
MeSH Terms: conditions — Premature Birth; Bronchopulmonary Dysplasia | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- nasal intermittent positive pressure ventilation group (Experimental)
  Interventions: Device: Nasal intermittent positive pressure ventilation (NIPPV); Device: lung ultrasound
- nasal continuous positive pressure ventilation group (Experimental)
  Interventions: Device: Nasal continuous positive airway pressure NCPAP; Device: lung ultrasound
- nasal high flow cannula group (Experimental)
  Interventions: Device: Nasal humidified heated high flow cannula (NHHHC); Device: lung ultrasound

INTERVENTIONS:
Device: Nasal humidified heated high flow cannula (NHHHC) — Patients in this arm will receive humidified heated high flow using Vapotherm device, USA. Stating with 2 L/min flow and increase gradually till 8L/minute, guided by oxygen requirements.
  Arms: nasal high flow cannula group
Device: Nasal intermittent positive pressure ventilation (NIPPV) — Patients in this arm will receive both PEEP (positive end expiratory pressure ) and PIP (peak inspiratory pressure) using SLE 5000/6000 device, UK . Pressures will be adjusted according to severity of respiratory distress.
  Arms: nasal intermittent positive pressure ventilation group
Device: Nasal continuous positive airway pressure NCPAP — Patients in this arm will receive PEEP (positive end expiratory pressure ), stating from 5 mbar to reach maximally 8 mbar.
  Arms: nasal continuous positive pressure ventilation group
Device: lung ultrasound — Lung ultrasound (LUS) machine is a mobile device (Philips HDll XE, USA) with s8-3 probe with a frequency range of 8-3 MHz will be used as ultrasound machine. Throughout the period of non-invasive respiratory support Patient will be monitored by: LUS,Heart rate, Respiratory rate, Mean arterial pressure, Oxygen saturation index, Oxygen index, PaO2, blood gases and Fractional inspired oxygen (Fio2).

SUMMARY:
This study aims to evaluate the effect of non-invasive ventilation (nIPPV)

, (nCPAP), and nasal high flow cannula (NHFC) as a primary mode of ventilation in preterm neonates <37 gestational week with moderate to severe RD using LUS as regard: I. Primary outcomes: Duration of non-Invasive ventilation. II. Secondary outcomes: Evaluation LUS over the 1 st 7 days of life or weaning from ventilation. Need for intubation and invasive ventilation. Duration of respiratory support. Need for surfactant. Oxygen saturation index and oxygen index. Broncho-pulmonary dysplasia; grade. Duration of hospital stay

ELIGIBILITY:
Inclusion Criteria: Preterm <37 wk. gestational age admitted to the NICU with spontaneous breathing and clinical manifestations of RD (tachypnea, nasal flaring, intercostal and subcostal retraction and or grunting).

Exclusion Criteria:

1. Obvious major congenital abnormalities.
2. Any of the baby intubated for resuscitation or for other reasons.
3. Neonates need invasive mechanical ventilation.
4. Pulmonary hemorrhage.
5. Severe cardiovascular instability.
6. Cardiopulmonary arrest needing prolonged resuscitation.
7. Birth asphyxia (one-minute Apgar score ≤ 3).
8. Major cardiac diseases (not including patent ductus arteriosus).

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-05-28 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of non-Invasive ventilation (NIV) | First two weeks of life.
  Describe the days of non-invasive ventilation , described in days number.

SECONDARY OUTCOMES:
Oxygen saturation index (OSI). | first one weeks of life.
  Mean airway pressure (MAP)X Fraction of inspired oxygen (FIO2) X SPO2 ( oxygen saturation) The score of OSI is recorded twice per day for first seven days.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Elshattbi hospital, Alexandria, Egypt